CLINICAL TRIAL: NCT02443896
Title: A Pilot Study to Investigate the Use of Pit and Fissure Sealants in Children Requiring Caries Related Dental Extractions Under a Chair General Anaesthetic
Brief Title: The Use of Pit and Fissure Sealants in Children Requiring Caries Related Dental Extractions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Birmingham Community Healthcare NHS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-089
Record Dates: First submitted 2015-04-01; First posted 2015-05-14 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2017-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sealant applied to molars (Experimental): All 'sealable' permanent molars will be sealed: Occlusal fissures and where appropriate, buccal pits (on lower molars) and palatal pits (on upper molars) will be sealed.
  If patient compliance is adequate, a resin based sealant will be used as the first choice material. The tooth is thoroughly cleaned, prepared with a special solution, and dried. The liquid sealant is then applied and allowed to set hard.
  Interventions: Procedure: Pit and Fissure Sealant of permanent molars
- No sealant applied to molars. (Sham Comparator): No molars will be sealed.
  Interventions: Procedure: No sealant of permanent molars

INTERVENTIONS:
Procedure: Pit and Fissure Sealant of permanent molars — The tooth is thoroughly cleaned, prepared with a special solution, and dried. The liquid sealant is then applied and allowed to set hard
  Arms: Sealant applied to molars
Procedure: No sealant of permanent molars — No sealant applied to permanent molars.
  Arms: No sealant applied to molars.

SUMMARY:
The purpose of thus study is to assess the feasibility and inform the planning of a proposed definitive randomised controlled clinical trial to investigate the efficacy of sealing permanent molars in children requiring caries related extractions under a chair General Anaesthetic.

DETAILED DESCRIPTION:
Objective:

To evaluate,

1. The ability to recruit based on failure to meet exclusion criteria, declining to participate or other reasons and retention rates based on subsequent withdrawals.
2. Feasibility and acceptability of placing sealants in this setting, based on compliance with the intervention.
3. Sealant retention rates based on the proportion of sealants that were fully intact, partially intact or lost after 24 months.
4. Two-year incidence of caries in permanent molars that were sound and suitable for sealants at the time of the pre-GA assessment, based on the proportion of children with:

   1. Experience of caries into dentine in at least one permanent molar
   2. Untreated caries into dentine in at least one permanent molar
5. Oral health related Quality of Life (OHRQoL) two years following caries related extractions under GA, based on the Child-Oral Impacts on Daily Performances (Child-OIDP) scale and separate questions relating to specified oral symptoms.
6. Oral health support provided by referring practitioners, within the 2 years following the dental GA, based on,

   1. Structured interview questionnaire to record parents' experience of preventive advice and treatment received, following the GA extractions
   2. Sealants identified at follow up that were not present at baseline or provided as part of the study

Recruitment and randomisation:

Recruitment was carried out over a total period of 8 months. However, during this time, the study investigator (AR) was only available to recruit participants on ad hoc dates. Therefore, to facilitate recruitment, referral letters were triaged to identify children that were likely to be eligible (based on age, postcode and reason for GA referral) so they could be scheduled on these dates.

Study information (including separate leaflets for parents and children) was posted a few weeks before the GA assessment appointment.

At this visit, clinicians responsible for completing the GA assessment, also screened children to identify those that had potentially sealable permanent molars, and they were then invited to see the investigator on the same day. Further to this, eligibility to take part in the study, based on the full list of inclusion criteria was confirmed following full verbal and written consent.

Results:

Although the recruitment period extended over 8 months, as explained earlier, the study investigator was only available to undertake enrolment on a limited number of ad hoc sessions throughout this time. Based on these, 132 children were assessed for eligibility.

ELIGIBILITY:
Inclusion criteria

* Children that are to have extraction of at least one carious tooth under a chair General Anaesthetic at Birmingham Dental Hospital
* Birmingham residents (as indicated by post code of home address)
* Be aged 5 to 15 years
* Be co-operative to a clinical dental examination
* Present with at least one permanent molar tooth that is 'sound and sealable'
* Be accompanied by an adult that has legal capacity to give informed consent

Exclusion criteria

Patients who at the pre-General Anaesthetic assessment visit present with:

* Signs of a systemic illness (e.g. coughs, 'colds', chicken pox) that might preclude placement of sealants
* Oral symptoms (e.g. pain, swelling) that would preclude sealant placement
* Parents unable to confirm (with a reasonable degree of certainty) that they would be contactable and able to attend for review during the 2 years duration of the study (e.g. because of plans to move)

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2017-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Caries incidence | 12 months
  The incidence of dental caries in permanent molars will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietrich, Principal Investigator — University of Birmingham
Locations (1):
- Birmingham Dental Hospital, Birmingham, United Kingdom